CLINICAL TRIAL: NCT01993264
Title: Standardization Of A Novel Method To Assess Fetal Cardiac Function: Myocardial Deformation Analysis
Brief Title: Fetal Cardiac Strain Imaging Research
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Ricardo H Pignatelli, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-33343
Record Dates: First submitted 2013-10-30; First posted 2013-11-25 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Myocardial Deformation
Keywords: Heart disease; Echocardiogram; Ultrasound; Heart defect; Heart Dysfunction; Pediatric Cardiologists; Prenatal
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Fetal Echocardiogram — Subjects will then have sequential, abbreviated fetal echocardiograms performed by designated, highly trained, and experienced sonographers every 4 weeks, from 20-36 weeks.

SUMMARY:
Cardiac disease in children may start early in life and evidence of cardiac disease can be seen during prenatal life. A variety of diseases diagnosed during fetal life can put children at risk for cardiac disease. The accurate assessment of cardiac function is important in these patients. A type of imaging scan called "fetal echocardiogram" is used to measure the contractility or squeeze of the heart. The fetal echocardiogram is a painless test and completely non-invasive.

This study aims to recruit women and fetuses to determine if this imaging scan can be used throughout the pregnancy to measure heart squeeze and develop normal values to help doctors better diagnose fetuses who may have cardiac disease before they are born.

DETAILED DESCRIPTION:
The subject will have to complete 6 fetal echocardiograms. A fetal echocardiogram is picture of the unborn baby's heart in motion made by bouncing sound waves off the heart and recording the echo. The procedure will be very similar to the ultrasounds that the subject is already receiving as part of her prenatal care.

The scans will start at week 20 of the subject's pregnancy and repeat every 3 weeks until week 38 of birth (whichever occurs first). The appointments will last approximately 30 minutes each and will be performed by one of two sonographers trained specifically in fetal echocardiography. One additional echocardiogram will be performed on the infant after birth, within the first two months of life. In addition to the scans, study staff will access the subject's medical record to collect information such as: age, ethnicity, race, medical history and health insurance status.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the obstetrics clinic at Texas Children's Hospital Pavilion for Women at the time of their second trimester screening ultrasound
* Fetus must have no recognizable disease at the second trimester screening ultrasound
* Willing to participate in a total of 5 fetal echocardiograms and one within 2 months after delivery
* English or Spanish literacy
* A four chamber view of the heart must be visible upon screening examination
* No fetal anatomic or growth abnormalities suspected on screening examination.

Exclusion Criteria:

* Subjects that meet the cutoff point for maternal obesity (BMI>30) and have identified risk factors for fetal cardiac dysfunction as determined by medical team.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients at the obstetrics clinic at Texas Children's Hospital Pavilion for Women at the time of their second trimester screening ultrasound will be asked to volunteer to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Inter-observer variability of institutional imaging and analysis protocol | 1 year
  Determine the inter-observer variability of our imaging and analysis protocol for the measurement of fetal myocardial deformation throughout gestation and after birth. The investigator will use the paired t-test to compare differences in measurement between the two observers at each time point.

SECONDARY OUTCOMES:
Normative reference ranges for various measures of myocardial deformation | 1 year
  Develop normative reference ranges for various measures of myocardial deformation (global left and right ventricular strain and strain rate) across gestation and after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Pignatelli, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States